CLINICAL TRIAL: NCT03622294
Title: A Clinical Analysis of Bella Blankets® Protective Coverlets Used to Increase the Image Quality of Mammograms, Aid as a Quality Standard for EQUIP Clinical Image Quality (CIQ) Compliance Measurements and Improve Patient Satisfaction.
Brief Title: A Clinical Analysis of Bella Blankets® Protective Coverlets
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beekley Medical (Industry)
Collaborators: Elizabeth Wende Breast Care, LLC (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 423-P-02
Record Dates: First submitted 2018-07-17; First posted 2018-08-09 (Actual); Last update posted 2019-06-27 (Actual); Status verified 2019-06

CONDITIONS: Screening Mammogram

STUDY DESIGN:
Intervention Model Description: Participants will be female, asymptomatic patients randomly scheduled for a screening mammogram.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Right Breast Mammogram Measurements and Survey (Experimental): A right breast screening mammogram will be performed with Bella Blankets protective coverlets on the imaging receptor plate, then removed from the equipment.
  The screening mammogram continues with a left breast and second right breast screening mammogram on a bare imaging receptor plate.
  Clinical image quality measurements for the right breast mammograms will automatically be captured by VolparaEnterprise for a comparative analysis.
  A patient satisfaction survey will be completed by each participant and the results will be analyzed.
  Interventions: Device: Bella Blankets protective coverlets

INTERVENTIONS:
Device: Bella Blankets protective coverlets — Bella Blankets protective coverlets is a Class II 510(k) Cleared (2008) single-use, adhering, non-woven fabric sheet applied to the mammography equipment receptor plate to provide a more comfortable mammogram.

SUMMARY:
This study will collect and compare clinical image quality measurements of randomly scheduled, asymptomatic, screening mammography patients, right breast mammogram performed with and without the use of Bella Blankets protective coverlets on the receptor plate.

The measurements will determine if the use of Bella Blankets protective coverlets increases the mammogram's clinical image quality and if Bella Blankets protective coverlets can be used as an aid for EQUIP compliance.

In addition, a patient satisfaction survey will be conducted with participants to determine if the use of Bella Blankets protective coverlets improves patient satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* Subject is Female of any race and ethnicity
* Subject is 40-75 years old
* Subject is scheduled for a screening mammogram
* Subject is willing and able to understand and read the Informed consent form
* Subject has been a patient at Elizabeth Wende Breast Care for 2 years or more

Exclusion Criteria:

* Subject is Male
* Subject has been a patient at Elizabeth Wende Breast Care for less than 2 years
* Subject has had a breast biopsy within the last 2 years
* Subject has had breast surgery within the last 2 years
* Subject is scheduled for a Diagnostic mammogram
* Subject suspects or may be pregnant
* Subject is currently pregnant or breastfeeding
* Subject has breast implants

Ages: 40 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 100 (Actual)
Dates: Start 2018-08-15 (Actual); Primary Completion 2018-11-06 (Actual); Study Completion 2019-06-25 (Actual)

PRIMARY OUTCOMES:
Clinical Image Quality (CIQ) Outcomes of a Participant's Right Breast Mammogram Performed with Bella Blankets Protective Coverlets on the Receptor Plate to a Bare Receptor Plate. | Through the completion of 100 participants; approximately 4 months
  Comparison of the Clinical Image Quality (CIQ) analytics, automatically captured by VolparaEnterprise, for the participant's right breast mammogram performed on a receptor plate with Bella Blankets protective coverlets to the same right breast mammogram performed on a bare receptor plate during the same screening mammogram visit.

SECONDARY OUTCOMES:
Patient Satisfaction Survey | Through the completion of 100 participants; approximately 4 months
  A questionnaire completed by the participant after their mammogram and prior to exit. The one-page questionnaire requires the participant answers each question by selecting one Likert Scale option about their experience with the use and without the use of Bella Blankets protective coverlets.

OTHER OUTCOMES:
Assessment as an Aid to Achieve Standards for Mammogram EQUIP Compliance Measurements. | At the completion of 100 participants; approximately 4 months from study initiation
  An assessment by the Principal Investigator,based on CIQ results and the FDA CIQ EQUIP standards, determining if Bella Blankets protective coverlets can be used by technologists to aid in achieving EQUIP compliance measurements in a mammogram.

CONTACTS AND LOCATIONS:
Locations (1):
- Elizabeth Wende Breast Care, LLC, Rochester, New York, United States